CLINICAL TRIAL: NCT02633150
Title: Assessing the Value of Red Grapes Polyphenol Supplementation on Metabolic Parameters in Obese Insulinoresistant Subjects : Study Randomized Versus Placebo
Brief Title: Assessing the Value of Red Grapes Polyphenol Supplementation on Metabolic Parameters in Obese Insulinoresistant Subjects
Acronym: POLYGIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9501; 2014-A01627-40 (Registry Identifier: ID RCB)
Record Dates: First submitted 2015-12-09; First posted 2015-12-17 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Obesity; Insulin Resistance; Menopause
Keywords: Obesity; insulinoresistant; menopausal women; polyphenol
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyphenol (Experimental): red grapes polyphenol supplementation on metabolic parameters in obese insulinoresistant subjects
  Interventions: Other: Supplementation with red grapes polyphenol
- Placebo (Placebo Comparator): Placebo supplementation on metabolic parameters in obese insulinoresistant subjects
  Interventions: Other: Supplementation with red grapes polyphenol

INTERVENTIONS:
Other: Supplementation with red grapes polyphenol

SUMMARY:
Obesity, chronic disease, is a real public health problem because of its high prevalence but also because of the high risk of complications, including insulin resistance (IR) and type 2 diabetes (T2D). The mechanisms involved in the development of IR are not well known. Oxidative stress and inflammation induced by food overload could be the initiators IR mechanisms in skeletal muscle, responsible for the use of nearly 80% glucose in response to insulin and therefore plays a major role in the regulation of glucose metabolism. Thus, an increase in ROS (Reactive Oxygen Species), markers of oxidative stress and chronic low-grade inflammation have been demonstrated in subjects with obesity, the latter decreasing in weight loss. Therapeutically, loosing weight is still very difficult these days, because of the complexity of this chronic disease. Thus, it is well established that restrictive diets to expose weight rebound, dramatic medically as in human terms for these patients. Support for physical activity is also difficult because of reduced mobility in patients, refer to the lack of motivation among some. Finally, investigators have no treatment "against-obesity" who have demonstrated a benefit / risk enough to be used routinely. It is therefore essential to seek other means of struggle against the IR, see help in weight loss.

In parallel, it is well established that the consumption of certain antioxidants, including polyphenols (PP) grape as extracts and whole foods, modulates favorably several pathways responsible for the development of IR in cell models animals. The results of antioxidants supplementation in humans are few and controversial. However, most supplementation studies in human used a PP, Resveratrol at supra nutritional doses (ie not compatible with a balanced diet of fruits and vegetables). In a previous study, investigators tested the interest of a supplementation with red grape PP nutritional doses in healthy subjects with metabolic risk (overweight subjects and related to the first degree of T2DM patients) on IR hyperinsulinemic euglycemic clamp measured. During this study, the PP have prevented the central mechanisms of muscle IR that are oxidative stress and mitochondrial dysfunction induced by a load fructose.

For this project, investigators propose to test the effect of a red grape PP supplementation at nutritional doses for 8 weeks on IR and weight loss in 30 obese insulin resistant. This is a double-blind randomized placebo-controlled. This supplementation will be associated with a standard support for their obesity performed routinely in the Nutrition and Diabetes unit.

Specific inclusion criteria: Female or male nondiabetic 50-65 years, BMI> 30 kg / m2 and with a HOMA> 3.

The main objective is to test whether supplementation PP improves systemic insulin sensitivity (GIR: rate glucose infusion) measured by hyperinsulinemic-euglycemic clamp (gold standard for measuring insulin sensitivity) in insulin-resistant obese subjects.

Secondary objectives are to:

* Test whether supplementation PP improves insulin sensitivity to tissue (fat and muscle) and compare the response to supplementation in these two tissues.
* Determining the cellular and molecular mechanisms involved in improving IR: regulation of inflammation, oxidative stress.
* Determine whether supplementation PP optimizes weight reduction compared to a standard single support.

NSN: The number of subjects required was evaluated from our previous work (2013 Hokayem et al.) Whose main objective was to assess the impact of PD versus placebo in first degree relatives of patients with diabetes type 2. Under a bilateral alternative hypothesis of a nonparametric test (Mann-Whitney), 1: 1 ratio, a power of 80% and an alpha risk of 0.05, the number of subjects was estimated at 15 per group.

Methodology: Anthropometric measurements, assessment of body composition (DEXA) system application characterization (metabolism, inflammation, oxidative stress, adipokines and insulin sensitivity: clamp hyperinsulinemic-euglycemic, lipopolysaccharides: LPS) / tissue characterization (biopsies of skeletal muscle and tissue adipose): insulin sensitivity, inflammation, oxidative stress, gene regulation (sirt1), mitochondrial activity / cell characterization (adipocyte precursor and muscle) insulin sensitivity, inflammation, oxidative stress, sirt1.

Investigators hope to demonstrate that a non-pharmacological treatment based on nutritional doses of PP supplementation can improve insulin sensitivity in insulin-resistant obese patients, refer to optimize weight loss compared to a standardized management of obesity and determine the mechanisms involved.

ELIGIBILITY:
Inclusion Criteria:

Specific inclusion criteria:

* Female or Male non diabetic
* Female postmenopausal, non hormono-substituted,
* 50-65 years,
* BMI> 30 kg / m2
* HOMA - IR > 3

Exclusion Criteria:

* active smoking, chronic inflammatory diseases, infection

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-10-06 (Actual); Primary Completion 2020-06-06 (Actual); Study Completion 2020-06-06 (Actual)

PRIMARY OUTCOMES:
Measure of systemic insulin sensitivity (estimated by GIR :rate glucose infusion) measured by hyperinsulinemic-euglycemic clamp | 8 weeks after supplementation
  GIR change after 8 weeks of supplementation

SECONDARY OUTCOMES:
Measure of insulin sensitivity to tissue (fat and muscle by measure ratio phosphoAKT/AKT measured by Western BLOT) before and after the supplementation | 8 weeks after supplementation
Measure of systemic concentration (by Multiplex) | 8 weeks after supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Ariane SULTAN, Pr, MD-PHD, Principal Investigator — Montpellier University Hospital
Locations (1):
- CHU Montpellier - Lapeyronie hospital, Montpellier, France